CLINICAL TRIAL: NCT02806323
Title: An Individually Tailored Yoga Program for the Treatment of Chronic Neck and Back Pain in a Low-income Population: A Feasibility Study
Brief Title: Individually Tailored Yoga Program for the Treatment of Chronic Neck and Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014-1582
Record Dates: First submitted 2016-05-03; First posted 2016-06-20 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Neck Pain Musculoskeletal; Back Pain, Unspecified
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Yoga Practice (Experimental): 12 week yoga intervention; 45 minutes/weekly practice Participants will be encouraged to practice their prescribed program of yoga at home, daily, for 20 minutes each day.
  Interventions: Other: Yoga practice

INTERVENTIONS:
Other: Yoga practice

SUMMARY:
The goal of this pilot study is to determine the feasibility of an individually tailored yoga program delivered in a group setting for the treatment of chronic neck and back pain in a low income population. Chronic pain is one of the most common, costly, and disabling conditions, and is often refractory to treatment. Yoga is a promising treatment for chronic pain. This pilot study will test the hypothesis that study subjects will participate in a voluntary 12 week yoga intervention for the treatment of chronic neck and back pain, as assessed by attendance at 12 weekly yoga practice sessions. Secondary outcomes will include change in pain and quality of life scores over the 12 week study period as assessed by the Visual Analog Scale for Pain Severity and EQ-5D-3L.

DETAILED DESCRIPTION:
This will be a pilot study involving only one group to assess the feasibility of an individually tailored program of yoga for the treatment of chronic neck and back pain. All study procedures will be completed in English and Spanish by study team members fluent in these languages, and using study materials printed in English and in Spanish. Potential participants will be recruited through flyers and referrals from providers at Wingra Family Medical Center. Interested potential participants will undergo screening in person or over the phone which will take approximately 15 minutes. If they are determined to be eligible, potential participants will meet with a member of the research team to receive information about the study and sign the consent form if they so choose. Consent will take approximately 15 minutes. Demographic information will be collected at the time consent is signed, this will take an additional 10 minutes. Following this, participants will have a 90 minute intake session with Adrienne Hampton, MD, RYT 200 [RYT 200 is the designation for a Registered Yoga Teacher with 200 hours of training] where the pain history will be elicited and the yoga program will be developed. Following this, participants will be encouraged to participate in the weekly drop-in practice sessions, where they will choose how much time they would like to spend asking questions, and receiving one on one practice instruction from Dr. Hampton. Participants will be encouraged to spend at least 45 minutes at the weekly practice session, which will include 10 minutes for completion of questionnaires. Participants will also be encouraged to practice their prescribed program of yoga at home, daily, for 20 minutes each day. The primary outcome measured will be attendance at yoga practice sessions. Additionally, indices of pain and quality of life will be assessed before, during, and after the study either in person or over the phone. Participants will also submit home yoga practice logs. All participants will be asked to complete a 30 minute exit interview in person at the end of the 12 week intervention period. The questionnaires are administered on paper, and participants will record their answers on paper. For the exit interview, the interviewer will read the questions to the participant, and then the interviewer will scribe on paper the participant's answers to the questions.Participants will be provided with bus passes to facilitate travel to study activities, and will be paid up to $50 for study participation.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will include neck and/or back pain on at least 5 days per week for >3 months, between ages 30-65, patient at Wingra family medical center, English or Spanish fluency.

Exclusion Criteria:

* Exclusion criteria will include regular yoga practice in the last 12 months, pregnancy, non-ambulatory, known metastatic lesions to bone, history of pathologic fracture, history of back or neck surgery in the past 6 weeks or planned in the next 6 months, psychotic mental health disorder, lack of decisional capacity, inability to adhere to proposed intervention and follow-up schedule.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Program feasibility based on participant attendance and practice logs | 12 weeks
  Feasibility of an individually tailored program of yoga for the treatment of chronic neck and/or back pain in a low-income population.

SECONDARY OUTCOMES:
Visual Analog Scale for Pain Severity | 12 weeks
  Visual Analog Scale for Pain Severity demonstrate positive relations to other self-report measures of pain intensity, to observed pain behavior and are sensitive to treatment effects.
EQ-5D™ (European Quality of Life) Instrument | 12 weeks
  EQ-5D™ is a standardized instrument for use as a measure of health outcome and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne Hampton, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Wingra Clinic, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided